CLINICAL TRIAL: NCT01047514
Title: Chronic Disease Self-Management Online Workshop for Canada
Brief Title: Healthier Living Canada
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: AHS Cancer Control Alberta (Other); National Council on Aging (NCOA) (Unknown)
Responsible Party: Principal Investigator, Kate Lorig, professor emertius, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SU-01052010-4604; 17832
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2013-04

CONDITIONS: Asthma; Chronic Disease
MeSH Terms: conditions — Asthma; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online Chronic Disease Self-management (Experimental): 6 week, online, small group online self-management workshop
  Interventions: Behavioral: Chronic Disease Self-Management Online Workshop

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Online Workshop — 6 week, online, small group self-management workshop
  Other Names: Healthy Living Canada

SUMMARY:
This study will evaluate the effectiveness of an online Chronic Disease Self-Management Program for participants in Canada living with chronic health conditions. This pilot will look for improvements in health status, health behaviors and health care utilization.

DETAILED DESCRIPTION:
The Healthier Living with Ongoing Health Problems online workshop provides self-management and self care skills training for people with long-term health conditions such as heart disease, lung disease, diabetes, multiple sclerosis, asthma and others. The workshop is delivered via the Internet over a six-week period. This is a pilot project, which means that it is being run for a limited time to test out its format and its usefulness for participants in Canada. A similar programme has been implemented in the USA, UK, and Australia, but it has to be tried now in Canada to see its usefulness for people in this country. .

The Online workshop is aimed at helping you to take better care of yourself and to better manage your health condition. It is hoped that at the end of the workshop you will be able to do the things you want to do and maintain the relationships that are important to you.

With the facilitators and other workshop participants, you will discuss:

* Dealing with fatigue/tiredness
* Dealing with difficult emotions
* Dealing with your physical symptoms
* Solving the problems caused by your condition
* Starting and maintaining an appropriate exercise or activity programme
* Managing medications
* Communicating better with health care professionals
* Communicating better with your friends, family and colleagues

ELIGIBILITY:
Inclusion Criteria:Adults 18 and over living with any chronic or long term health condition such as heart disease, lung disease, diabetes. Exclusion Criteria:Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
health behaviors | 6 month and 1 year
health utilization | 6 month and 1 year
health status | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States